CLINICAL TRIAL: NCT05470608
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Single-Ascending Dose Escalation Study to Assess the Safety and Efficacy of SL-1002 Injectable for Treatment of Knee Pain Associated With Osteoarthritis
Brief Title: Phase II Study to Assess Safety and Efficacy of SL-1002 for Osteoarthritic Knee Pain
Acronym: COMPASS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Saol Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1010-01
Record Dates: First submitted 2022-07-20; First posted 2022-07-22 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Osteoarthritis, Knee Pain
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SL-1002 (Experimental): SL-1002 injectable solution, single dose
  Interventions: Drug: SL-1002
- Matching placebo (Placebo Comparator): Matching placebo injectable solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SL-1002 — SL-1002 injectable solution
  Arms: SL-1002
Drug: Placebo — Matching placebo injectable solution
  Arms: Matching placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, single ascending dose escalation study to assess the safety and efficacy of single treatment exposure of an injectable formulation of SL-1002 for the treatment of knee pain associated with osteoarthritis. Phase A of the study will enroll 3 cohorts of 8 patients per cohort, for a total of 24 patients. Patients will be randomized to receive either SL-1002 or placebo in a 3:1 ratio within each given cohort. Phase B of the study will enroll a minimum of 92 up to a maximum of 108 patients. Patients will be randomized to receive either SL-1002 or placebo in a 3:1 ratio at the recommended dose determined from Phase A. The study period will be up to 168 days inclusive of a screening period of up to 28 days.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients 35 years of age or older, with a Body Mass Index (BMI) of 18.0 to 40.0 kg/m2 and a total body weight of ≥50.0 kg for males and ≥45.5 kg for females.
2. Patients with chronic knee pain resulting from osteoarthritis for greater than 6 months prior to study Screening Visit 1 that interferes with functional activities (e.g., ambulation, prolonged standing, etc.).
3. Patients currently experiencing continued pain despite receiving at least 3 months of conservative treatments, inclusive of activity modification, home exercise, protective weight bearing, and/or use of analgesics (e.g., acetaminophen or NSAIDs).
4. Patients with a baseline average pain score of ≥ 6 on an 11-point NRS scale as "usual level of pain over the past 24 hours during weight-bearing activities" for the index knee at Screening. The baseline average pain score is computed by finding the mean of the daily NRS pain intensity scores reported during the 7-day run in period.
5. Patients with Kellgren-Lawrence Grade 2 (mild) or Grade 3 (moderate) radiologically confirmed osteoarthritis (via x-ray/MRI/CT) within 6 months of study Screening Visit 1.
6. Patients with a baseline Knee Injury and Osteoarthritis Outcome Score (KOOS) pain subscale score ≥ 19 and ≤ 67 in the index knee.
7. Patients taking analgesics, inclusive of membrane stabilizers (e.g., Neurontin/gabapentin) and/or antidepressants (e.g., Cymbalta/duloxetine), for osteoarthritis associated knee pain must be on a stable dose for at least 6 weeks prior to study Screening Visit 1. Patients must agree to not alter the dose of analgesics for the duration of the study without prior approval from the Investigator.
8. Female patients of childbearing potential who are sexually active with a male partner must be willing to use one of the following acceptable contraceptive methods throughout the study and for 30 days after the last study drug administration:

   1. Intra-uterine contraceptive device placed at least 4 weeks prior to study drug administration;
   2. Male condom with intravaginally applied spermicide starting at least 21 days prior to study drug administration;
   3. Hormonal contraceptives starting at least 4 weeks prior to study drug administration must agree to use the same hormonal contraceptive throughout the study;
   4. Sterile male partner (vasectomized since at least 6 months).
9. Female patients of non-childbearing potential as defined below:

   1. Postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) and estradiol levels consistent with menopause).
   2. Pre-menopausal females with one of the following:

      * Documented tubal ligation
      * Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion
      * Hysterectomy
      * Documented bilateral oophorectomy.
10. Patients must agree to see one treating physician (study Investigator) for knee pain treatment for study duration.
11. Patients who have a positive response to a single genicular nerve block of the index knee using 1.5 - 3mL of lidocaine 2% solution administration to the genicular nerves planned for treatment in each cohort (0.5mL per nerve). A positive response to the qualifying lidocaine prognostic block is defined as ≥ 80% pain reduction within 60 minutes of receiving the lidocaine injections and ≥ 80% pain relief for a duration of at least 60 minutes as documented on a standardized 6-hour pain log.
12. Patients must be able to understand and be able to complete all assessments associated with the study outcome measures.
13. Patients must be able to understand the informed consent and be willing to provide written informed consent. Patients must be able to comply with the requirements of the protocol for the entire duration of the study.

Exclusion Criteria:

1. Patients with evidence of inflammatory arthritis (e.g., rheumatoid arthritis) or any other systemic inflammatory condition (e.g., gout, pseudogout). 2. Current diagnosis of fibromyalgia. 3. Patients with evidence of neuropathic pain affecting the index knee. 4. Patients with prior or planned lower limb amputation. 5. Patients who have received an intra-articular steroid injection into the index knee within 90 days of study Screening Visit 1. 6. Patients who have received hyaluronic acid injection, Platelet Rich Plasma (PRP), stem cell or arthroscopic debridement/lavage injection into the index knee within 180 days of study Screening Visit

* Patients who have received prior radiofrequency ablation or any other neurolytic procedure of the genicular nerves of the index knee within 1 year of study Screening Visit 1.
* Patients who have received prior partial, resurfacing, or total knee arthroplasty of the index knee (residual hardware).
* Patients with clinically significant ligamentous laxity of the index knee as per Investigator discretion.
* Patients with clinically significant valgus/varus deformities or evidence of pathology (other than osteoarthritis of the knee) that materially affects gait or function of the index knee or is the underlying cause of the knee pain and/or functional limitations.
* Patients who are extremely thin and those with minimal subcutaneous tissue thickness that could place the patient at risk of a chemical skin burn, at the discretion of the Investigator.
* Patients with a pending or active compensation claim, litigation or disability remuneration (possibility of secondary gain).
* Patients with chronic pain associated with significant psychosocial dysfunction.
* Patients with a Patient Health Questionnaire - 9 (PHQ-9) score of >10 (indicative of a state of moderate depression).
* Patients with a systemic infection, active joint infection, or localized infection at the planned needle entry sites (patient may be considered for inclusion once infection is resolved).
* Patients with history of uncontrolled coagulopathy or unexplained or uncontrollable bleeding that cannot be corrected, and patients with coagulopathy or who are being treated with anticoagulants.
* Patients with moderate to severe hepatic impairment or moderate to severe renal impairment.
* Identifiable anatomical variability that would materially alter the procedure as described in the protocol.
* Patients currently prescribed opioid medications at a dose of >50 daily morphine equivalents.
* Patients with uncontrolled immunosuppression (e.g., AIDs, cancer, diabetes) as per Investigator discretion.
* Female patients who are pregnant or planning to become pregnant during the duration of the study.
* Female patients who are breast-feeding.
* Patients who are unable or unwilling to comply with the requirements of the protocol.
* Patients taking any of the following concurrent medications/over-the counter products (refer to Appendix 8 in full protocol for a list of applicable medications): c. Probenecid or other organic anion transporter (OAT3) inhibitors. d. Inhibitors of CYP2E1, such as disulfiram.
* Patients with known allergies or hypersensitivity to iodinated contrast medium and gadolinium-based contrast medium. Known allergies or hypersensitivity to phenol and/or lidocaine and/or their excipients.
* Patients with a documented history or evidence of alcohol or drug abuse within 1 year of study screening visit 1.
* Participation in a clinical research study involving the administration of an investigational or marketed drug or device within 30 days of study Screening Visit 1, administration of a biological product in the context of a clinical research study within 90 days prior to the first dosing, or concomitant participation in an investigational study involving no drug or device administration.
* Patients with clinically significant ECG abnormalities or vital sign abnormalities at during study Screening Visit 1. Patients with ECG or vital sign abnormalities deemed nonclinically significant or unlikely to result in clinical compromise by the Principal Investigator may be considered for study inclusion.
* Patients with clinically significant laboratory results (as judged by the Principal Investigator).
* Any condition, in the opinion of the Principal Investigator, that may pose a significant risk to the patient, confound the results of the study or interfere significantly with the patient's participation in the study.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2022-06-13 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of treatment emergent adverse events (TEAEs) overall | Time of study drug administration to end of study visit (day 168)
  TEAE timepoints will be observed from the time point of administration of total dose until end of study visit (day 168)
Improvement of knee pain | Change from baseline to Month 3 in 11 point NRS score
  Change in weekly average daily pain intensity via Numeric Rating Scale (NRS) score at Month 3

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Denver Spine & Pain Institute, Greenwood Village, Colorado
  - International Spine, Pain & Performance Center, Washington D.C., District of Columbia
  - Prime Medical Research, Coral Gables, Florida
  - Conquest Research, Winter Park, Florida
  - Northwestern University, Chicago, Illinois
  - Mayo Clinic, Rochester, Minnesota
  - Cooper Neurological Institute, Camden, New Jersey
  - Center for Clinical Research, Winston-Salem, North Carolina
  - Pacific Sports and Spine, Eugene, Oregon
  - University Orthopedics Center, Altoona, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Institute of Precision Pain Medicine, Corpus Christi, Texas
  - Precision Spine Care, Tyler, Texas
  - University of Utah School of Medicine, Salt Lake City, Utah
  - Virginia iSpine Physicians, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No